CLINICAL TRIAL: NCT00975520
Title: A Randomised Trial of Post-operative Radiation Therapy Following Wide Excision of Neurotropic Melanoma of the Head and Neck
Brief Title: Neurotropic Melanoma of the Head and Neck
Acronym: RTN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01.09; 2009/039 (Other: HREC); ACTRN12610000478011 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Melanoma
Keywords: Neurotropic; Melanoma; Observation; Radiation Therapy; Relapse
MeSH Terms: conditions — Melanoma; Recurrence | interventions — Observation; Surgical Procedures, Operative; Radiotherapy; Radiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiation Therapy (Active Comparator): Investigational Treatment
  Interventions: Radiation: Radiation Therapy
- Observation (Other): Observation
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Patients will be observed after surgery until recurrence when they will be offered radiation therapy
  Other Names: Surgery Alone
  Arms: Observation
Radiation: Radiation Therapy — Patients randomised to the Investigational treatment arm, will receive adjuvant curative post-operative radiation therapy aiming to reduce the rate of local recurrence. The recommended dose prescribed is 48 Gy in 20 fractions over 4 weeks.
  Other Names: RT, radiotherapy
  Arms: Radiation Therapy

SUMMARY:
This is a 2-armed randomised controlled trial comparing surgery alone with surgery plus post-operative radiation therapy for patients with completely resected primary melanoma showing histological features of neurotropism. Uncontrolled studies suggest that this form of primary melanoma has a high risk of local recurrence and that postoperative radiation therapy may substantially reduce that risk. Patients who are eligible on the basis of the pathology of the excised melanoma will be offered the opportunity to take part in the trial. Those randomised to receive radiation therapy will be treated with a simple technique encompassing the surgical bed plus a margin. Radiation will commence within 3 months of surgery (maximum of 14 weeks from surgery to start of radiotherapy).

DETAILED DESCRIPTION:
Background Melanoma is a serious and common malignancy in Australia. It is the third most common cancer in Australia and approximately 1000 Australians will die of the disease each year.At least a quarter of these will be patients under the age of 40 years.

Neurotropism, defined as invasion by melanoma of peripheral neural tissue, is a feature of the disease that may predispose towards a high local recurrence rate. Local recurrence, particularly in the head and neck region often requires more extensive, potentially morbid surgery. Neurotropism is especially likely to occur in desmoplastic melanoma where it may be as high as 40 - 60%.6-8 Desmoplastic melanoma tends to occur in a slightly older age group than conventional types of melanoma and most often occurs in the head and neck region in individuals with chronic sun damage.

The management of localised neurotropic melanoma has traditionally been with surgery. Recommendations are that surgical margins should be at least 2 cm.There are some patients where this margin is not achievable due to the location of the tumour close to important anatomical structures. Uncontrolled studies suggest that radiation therapy may reduce the risk of local recurrence in those patients although there are no randomised trials to confirm this hypothesis.

Postoperative adjuvant radiation therapy has been shown in a randomised trial led from Australia, to reduce regional recurrence rates in nodal melanoma.There are no previously conducted randomised controlled trials addressing a similar question for neurotropic melanoma. The only reports are in relation to retrospective reviews that suggest a benefit for postoperative radiation therapy after surgery. It is unlikely that this trial will be done outside of Australia.

Hypotheses

1. Radiation therapy after surgery for neurotropic melanoma improves local control.
2. This can be achieved without a significant increase in treatment morbidity or reduction in quality of life.

Primary Objective

• To determine, in patients who have undergone surgery with curative intent for neurotropic melanoma, whether there is a difference in the rate and timing of local (in field) recurrence between patients who are treated with post-operative radiation therapy and those that are initially observed.

Secondary Objectives

* To determine, in these patients, whether there is a difference in progression-free survival, patterns of relapse and overall survival between patients treated with surgery alone and those treated by surgery plus adjuvant radiation therapy.
* To determine, in these patients, whether there is a difference in morbidity and quality of life between patients treated with surgery alone and those treated with surgery plus adjuvant radiation therapy

Methodology This is a 2-armed randomised controlled trial comparing surgery alone with surgery plus post-operative radiation therapy for patients with completely resected primary melanoma showing histological features of neurotropism. Patients who are eligible on the basis of the pathology of the completely excised melanoma will be offered the opportunity to take part in the trial. Those randomised to receive radiation therapy will be treated with a simple technique encompassing the surgical bed plus a margin within 3 months of surgery. The same regimen which was used in the nodal trial will be used in this study. Patients in the observation arm who subsequently recur in field may be offered further surgery followed by radiation therapy.

Randomisation Methods Patients will be randomised in the ratio of 1:1 between the two arms, radiation therapy and no radiation therapy. Allocation to the treatment arm will be stratified by institution and tumour site (head or neck) using randomly permuted blocks. Patients who are eligible on the basis of their pathology of excised melanoma will be offered the opportunity to take part in the trial. While males and females will both be considered equally for participation on the trial, there is no way of knowing if the ratio will be 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Has provided written informed consent for participation in this trial
* Histologically confirmed neurotropic primary melanoma

  * Neurotropism is identified pathologically by the presence of melanoma cells around nerve sheaths (perineural invasion) or within nerves (intraneural invasion).
  * Occasionally, the tumour itself may form neuroid structures (termed 'neural transformation'; this is also regarded as neurotropism)
  * "normal"-looking nerves that appear to be "entrapped" within the tumour should not be regarded as neurotropism
* Tumour located above the clavicle and below the jaw or occiput (neck primary) or above the jaw/occiput (head primary)
* Complete macroscopic resection of all known disease
* No previous surgery for melanoma (other than complete macroscopic resection as stated above)(i.e. Not recurrent disease)
* No evidence of in-transit, nodal or distant metastases as determined by clinical examination, CT or MRI
* ECOG performance status score of 2 or less
* Life expectancy greater than 6 months
* Patients capable of childbearing are using adequate contraception
* Available for follow up

Exclusion Criteria:

* Women who are pregnant or lactating
* Intercurrent illness that will interfere with the radiation therapy such as immunosuppression due to medication or medical condition
* Clinical and/or MRI evidence of a named cranial or cervical nerve involvement by tumour
* Inability to localise surgical bed on CT scans and/or surgical margins (cm) not known
* Previous radical radiation therapy to the head and neck, excluding superficial radiation therapy to cutaneous SCC or basal cell carcinoma, which is not within or overlapping the tumour bed
* High risk for poor compliance with therapy or follow-up as assessed by investigator
* Patients with prior cancers, except: those diagnosed ≥ 5 years ago with no evidence of disease relapse and clinical expectation of relapse of less than 5%; prior successfully treated Level 1 cutaneous melanomas ≥ 2 years ago; or non-melanoma skin cancer; or carcinoma in situ of the cervix
* Albinism
* Participation in other clinical trials with the same primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2021-01 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Time to local relapse | 5 years from the date of randomisation

SECONDARY OUTCOMES:
Relapse free survival | 5 years from date of randomisation
Time to Relapse | 5 years from date of randomisation
Overall survival | 5 years from date of randomisation
Cancer specific survival | 5 years from date of randomisation
Patterns of relapse | 5 years from date of randomisation
Late Toxicity | 5 years from date of randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Foote, Study Chair — Princess Alexandra Hospital
Locations (16):
- United States (2):
  - Memorial Sloan Ketttering, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Australia (13):
  - Calvary Mater Hospital, Newcastle, New South Wales
  - Melanoma Institute Australia / Royal Prince Alfred Hospital, North Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Radiation Oncology Services - Mater Centre, South Brisbane, Queensland
  - Radiation Oncology Queensland (ROQ), Toowoomba, Queensland
  - Townsville Cancer Centre, Townsville, Queensland
  - Genesis Care: Tugun, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Norfolk and Norwich University Hosptial, NHS Foundation Trust, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not sharing IPD

REFERENCES:
- See also: Please visit this website for further trial specific information — https://www.masc.org.au/